CLINICAL TRIAL: NCT00587405
Title: Prospective Randomized Study of Cryotherapy Versus Argon Plasma Coagulation Therapy for Treatment Of Watermelon Stomach
Brief Title: Cyrotherapy vs. APC in GAVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Louis-Michel Wong Kee Song, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2261-05
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2010-04

CONDITIONS: Watermelon Stomach
Keywords: Watermelon Stomach; Cryotherapy; Argon Plasma Coagulation
MeSH Terms: conditions — Gastric Antral Vascular Ectasia | interventions — Cryotherapy; Argon Plasma Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Cryotherapy
  Interventions: Procedure: cryotherapy
- 2 (Active Comparator): Argon Plasma Coagulation
  Interventions: Procedure: Argon Plasma Coagulation

INTERVENTIONS:
Procedure: cryotherapy — The Polar Wand device (GI Supply, Wayne, PA) is FDA 510(k) approved for endoscopic tissue ablation in the GI tract. It consists of a portable cryogen-containing unit and a single-use flexible cryogen spray catheter, designed for use with CO2 that is supplied in standard 20-lb cylinders. Controlled delivery of the cryogen is achieved by a foot pedal, and the tip of the catheter is maintained at about 1 cm from the mucosa. A cryogenic spray is applied to all vascular lesions until a whitened appearance of the mucosa is achieved within 3-5 seconds. Affected areas will be 'painted' by the spray catheter starting at the pylorus and sweeping proximally.
  A proton pump inhibitor, at double dose, will be prescribed for 1 month after each APC or cryotherapy session to promote mucosal healing post therapy.
  Arms: 1
Procedure: Argon Plasma Coagulation — As per current clinical standard, the APC 300 device (ERBE Inc., Marietta, GA) will be used in this study. Targeted ablation of all vascular ectasias as best possible will be performed in standard fashion using an end-firing probe at a setting of 60 W and 2 L/min argon flow rate.A proton pump inhibitor, at double dose, will be prescribed for 1 month after each APC or cryotherapy session to promote mucosal healing post therapy
  Arms: 2

SUMMARY:
To see if either method of treatment for Watermelon Stomach shows better results

DETAILED DESCRIPTION:
Watermelon stomach (WS) is endoscopically recognized by characteristic stripes of angioectasias involving primarily the antrum, and causes transfusion-dependent anemia in the majority of patients. Current endoscopic treatment options, including argon plasma coagulation (APC) Endoscopic cryotherapy is a novel technique that has the potential to safely and more effectively treat WS by virtue of its mechanism of injury and mode of application.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed WS at endoscopy that is associated with significant anemia (Hb < 10 g/dl) and/or overt bleeding (melena, hematochezia or hematemesis) and/or blood transfusions within the past 6 months
2. Able to give informed consent
3. Age > 18 years

Exclusion Criteria:

1. Endoscopic or histological findings inconsistent with WS
2. Known coagulopathy (INR > 2), severe thrombocytopenia (platelet count < 50,000), or bleeding diathesis
3. Endoscopic treatment of WS within the past month
4. Unable or unwilling to give informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
the proportion of clinical responders (no overt and hematological evidence of ongoing bleeding) and non-responders | 6 months

SECONDARY OUTCOMES:
Endoscopic response will constitute the secondary outcome | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Louis M Wongkeesong, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo CLinic, Rochester, Minnesota, United States